CLINICAL TRIAL: NCT04224636
Title: A Randomized, 2-arm Non-comparative Phase II Study on the Efficacy of Atezolizumab and Roche Bevacizumab (Atezo/Bev) Followed by On-demand Selective TACE (sdTACE) Upon Detection of Disease Progression or of Initial Synchronous Treatment With TACE and Atezo/Bev on 24-months Survival Rate in the Treatment of Unresectable Hepatocellular Carcinoma Patients
Brief Title: Atezolizumab/Bevacizumab Followed by On-demand TACE or Initial Synchronous Treatment With TACE and Atezolizumab/Bevacizumab
Acronym: DEMAND
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Enrico De Toni, Professor, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-HEP-0418; 2019-002430-36 (EudraCT Number)
Record Dates: First submitted 2019-12-19; First posted 2020-01-13 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma Non-resectable
MeSH Terms: interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Up-front Atezo/Bev, then TACE (Experimental): Patients will receive atezolizumab and bevacizumab iv every three weeks for up to 24 months. Upon detection of at least one unequivocal progressive hepatic lesion, selective TACE directed against progressive lesion(s) (sdTACE) will be performed. RFA or MWA are permitted as alternative to TACE to treat one or more lesion that cannot be reasonably selectively targeted by TACE
  Interventions: Combination Product: Atezolizumab Injection, Bevacizumab Injection
- Atezo/Bev combined with TACE (Experimental): First TACE will be performed as selectively as possible against all viable tumor lesions. Atezo/Bev will be initiated within three days from TACE. Upon detection of at least one unequivocal progressive hepatic lesion, treatment with Atezo/Bev will be continued if RFA or MWA can be used to treat this/these progressive lesion.
  Interventions: Combination Product: Atezolizumab Injection, Bevacizumab Injection

INTERVENTIONS:
Combination Product: Atezolizumab Injection, Bevacizumab Injection — Atezolizumab and Bevacizumab will be administered prior to or in combination with TACE
  Other Names: Chemoembolisation (TACE)

SUMMARY:
Aim of the study is to evaluate the efficacy of up-front atezolizumab/ bevacizumab (Atezo/Bev) followed by on-demand selective transarterial chemoembolization (sdTACE) and of initial synchronous treatment with TACE and Atezo/Bev in the treatment of unresectable HCC patients.

ELIGIBILITY:
Key Inclusion Criteria

1. Patient's signed informed consent
2. Age ≥18 years at time of signing Informed Consent Form
3. Ability to comply with the study protocol, according to investigator's judgement
4. Life expectancy of at least 12 weeks
5. HCC with histologically confirmed diagnosis
6. Disease that is not amenable to curative surgical and/or local ablation but eligible for TACE
7. ECOG Performance Status of 0 or 1
8. Child-Pugh class A or B7
9. Adequate hematologic and end-organ function
10. Negative HIV test at screening

Key Exclusion Criteria

1. Diffuse HCC or presence of vascular invasion or extrahepatic spread or more than 7 lesions or at least one lesion >= 7 cm
2. Clinically relevant ascites
3. Uncontrolled pleural effusion or pericardial effusion
4. History or presence of hepatic encephalopathy
5. Co-infection of HBV and HCV
6. Patients on a liver transplantation list.
7. Prior systemic therapy for HCC
8. Prior treatment with TACE or selective internal radiation treatment (SIRT)
9. Any condition representing a contraindication to TACE
10. Major gastrointestinal bleeding within 4 weeks prior to randomization, untreated or incompletely treated varices with bleeding or high-risk for bleeding.
11. Active or history of autoimmune disease or immune deficiency
12. Prior allogeneic stem cell or solid organ transplantation
13. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
14. Active tuberculosis
15. Severe infection requiring antibiotics within 4 weeks prior to randomization
16. Significant cardiovascular disease
17. History of congenital long QT syndrome or corrected QT interval >500 ms at screening ECG
18. Inadequately controlled arterial hypertension or prior history of hypertensive crisis or hypertensive encephalopathy
19. Significant vascular disease including aortic aneurysm requiring surgical repair or peripheral arterial thrombosis with 6 months prior to randomization
20. History of abdominal or tracheoesophageal fistula or gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to randomization.
21. History or clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding. Evidence of abdominal free air that is not explained by paracentesis or recent surgical procedure
22. History of intra-abdominal inflammatory process within 6 months prior to randomization, including but not limited to peptic ulcer disease, diverticulitis, or colitis
23. Evidence of bleeding diathesis or significant coagulopathy
24. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
25. Uncontrolled tumor-related pain. Patients requiring pain medication must be on a stable regimen at enrollment.
26. Severe, non healing or dehisced wound, active ulcer, or untreated bone fracture
27. History of malignancy other than HCC, with the exception of patients who have been disease-free for at least five years before enrollment or patients with adequately treated and completely resected basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer, stage I uterine cancer
28. Current or recent (within 10 days of randomization) use of acetylsalicyclic acid or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol
29. Current or recent (within 10 days prior to randomization) use of full dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purpose.
30. Chronic daily treatment with a nonsteroidal anti-inflammatory drug (NSAID). Occasional use of NSAIDs for the symptomatic relief of medical conditions such as headache or fever is allowed.
31. Treatment with a live, attenuated vaccine within 4 weeks prior to randomization, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the last dose of atezolizumab
32. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and antiPD-L1 therapeutic antibodies
33. Hypersensitivity to atezolizumab or bevacizumab or any of the excipients, known hypersensitivity to Chinese hamster ovary cell products, known hypersensitivity to human or humanized antibodies
34. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to randomization
35. Treatment with systemic immunosuppressive medication within 2 weeks prior to randomization, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible.

    Inhaled corticosteroids for chronic obstructive pulmonary disease or bronchial asthma, supplemental mineralocorticosteroids or low-dose corticosteroids for adrenalcortical insufficiency are allowed.
36. Major surgical procedure other than for diagnosis, open biopsy, or significant traumatic injury within 28 days prior to randomization, or abdominal surgery, abdominal interventions or significant abdominal traumatic injury within 60 days prior to randomization or anticipation of need for major surgical procedure during the course of the study or non-recovery from side effects of any such procedure
37. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 3 days prior to the first dose of bevacizumab
38. Pregnant or breastfeeding females
39. Participation in a clinical trial or experimental drug treatment within 28 days prior to inclusion in the clinical trial or within a period of 5 half-lives of the substances administered in a clinical trial or during an experimental drug treatment prior to inclusion in the clinical trial, depending on which period is longest, or simultaneous participation in another clinical trial while taking part in this clinical trial.
40. Patient committed to an institution by virtue of an order issued either by the judicial or the administrative authorities
41. Patient possibly dependent from the investigator including the spouse, children and close relatives of any investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 24 months
  Response is defined by RECIST 1.1 and mRECIST

SECONDARY OUTCOMES:
Median overall survival (mOS) | 24 months
  Defined as the time from treatment initiation until death
Progression-free survival (PFS) | 24 months
  Progression is defined according RECIST 1.1 and mRECIST
24-months survival rate | 24 months
  Percentage of patients alive after 24 months since randomization
Complete response rate (CRR) | 24 months
  Defined by the percentage of patients with disappearance of tumor manifestation at radiological evaluation
Disease control rate (DCR) | 24 months
  Defined as the percentage of patients who have achieved complete response, partial response and stable disease
Time to deterioration of liver function | 24 months
  Defined as time from randomization to worsening of CTCAE grade for any of these parameters: aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, albumin, and international normalized ratio (INR)
Time to untreatable progression | 24 months
  defined as time from randomization to progression not amenable to local treatment as per protocol, occurrence of vascular invasion or of extrahepatic spread, worsening of liver function to Child-Pugh score 8 or higher
Time to stage-progression | 24 months
  Defined as time from randomization to disease progression to BCLC C stage
Time to first TACE (arm A) | 24 months
  Defined as time from randomization to disease to the first TACE
Quality of life (QOL) | 24 months
  Standardized assessment will be performed by using EORTC QLQ-C30 - European Organisation for Research and Treatment of Cancer - Quality of Life Core Questionnaire 30 items
Quality of life (QOL) | 24 months
  Standardized assessment will be performed by using EORTC QLQ-HCC18 - European Organisation for Research and Treatment of Cancer - Quality of Life Core Questionnaire - Hepatocellular carcinoma module 18
Adverse Events | 24 months
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (7):
- Germany (7):
  - University of Bonn, Bonn
  - University Hospital Cologne, Cologne
  - Hospital of the University of Munich, Munich
  - Klinikum Rechts der Isar of the Technical University Munich, Munich
  - University Hospital Regensburg, Regensburg
  - University Hospital Tübingen, Tübingen
  - Würzburg University Hospital, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Toni EN. Immune checkpoint inhibitors: use them early, combined and instead of TACE? Gut. 2020 Oct;69(10):1887-1888. doi: 10.1136/gutjnl-2019-319658. Epub 2019 Oct 14. No abstract available. PMID 31611301
- [Derived] Ben Khaled N, Seidensticker M, Ricke J, Mayerle J, Oehrle B, Rossler D, Teupser D, Ehmer U, Bitzer M, Waldschmidt D, Fuchs M, Reuken PA, Lange CM, Wege H, Kandulski A, Dechene A, Venerito M, Berres ML, Luedde T, Kubisch I, Reiter FP, De Toni EN. Atezolizumab and bevacizumab with transarterial chemoembolization in hepatocellular carcinoma: the DEMAND trial protocol. Future Oncol. 2022 Apr;18(12):1423-1435. doi: 10.2217/fon-2021-1261. Epub 2022 Jan 27. PMID 35081747